CLINICAL TRIAL: NCT07009418
Title: Coronary Computed Tomography Angiography Versus Standard Care in High-Risk Patients After Percutaneous Coronary Intervention
Brief Title: Smart Angioplasty Research Team-Coronary CT Angiography Versus Standard Care as Follow-up Strategies in High-Risk Patients After PCI (SMART-CARE)
Acronym: SMART-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC19801001
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary intervention; coronary computed tomography angiography; follow-up strategy
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Pragmatic, prospective, multi-center, open label, randomized controlled, superiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participant and care provider cannot be blinded. But, investigator and clinical outcoem assessor will be blinded about the randomly allocated groups. Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surveillance by CCTA Strategy Group (Experimental): In the surveillance by CCTA group, patients will be evaluated by CCTA at 1 year from index hospitalization. CCTA will be done according to current acquisition guidelines.
  Interventions: Diagnostic Test: Coronary CT Angiography (CCTA)
- Standard Care Strategy Group (No Intervention): In the standard care group, patients will be managed according to the current guidelines. Regardless of symptoms, periodic visits will be performed by the charged physician. Secondary prevention including cardiovascular risk factor control, assessment of disease status, and comorbidities, and GDMT will be meticulously performed. In patients without a change in clinical or functional status, further evaluation by CCTA or non-invasive functional tests will not be performed. In this group, CCTA or non-invasive functional tests will be performed only for patients with significant change in clinical or functional status or with symptoms refractory to medical treatment.6,8 Whether patients will be referred for invasive coronary angiography will be determined by the charged physician according to patient's clinical or functional status and the results from CCTA or non-invasive functional tests according to current guidelines.

INTERVENTIONS:
Diagnostic Test: Coronary CT Angiography (CCTA) — In the surveillance by CCTA group, patients will be evaluated by CCTA at 1 year from index hospitalization. CCTA will be done according to current acquisition guidelines. Downstream management according to the results from CCTA will be performed under recommendations from current guidelines.
  Arms: Surveillance by CCTA Strategy Group

SUMMARY:
The aim of the SMART-CARE trial is to compare clinical outcomes between coronary CT angiography (CCTA) versus standard care as follow-up strategies in high-risk patients after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Advancements in drug-eluting stents, physiology-guided treatment decisions, intravascular imaging-guided procedural optimization, and adjunctive medical therapy have significantly improved prognosis after percutaneous coronary intervention (PCI). However, high-risk patients-particularly those with complex coronary artery lesions or high-risk clinical conditions such as acute myocardial infarction with or without cardiogenic shock at presentation, diabetes mellitus which requires medical treatment (oral hypoglycemic agents or insulin), end-stage renal disease under dialysis, or multi-vascular disease-continue to have a significantly higher risk of adverse cardiovascular events. In this regard, meticulous follow-up, including periodic assessment of clinical and functional status, guideline-directed medical therapy (GDMT), and secondary prevention strategies are important, and current guidelines strongly recommend these measures as a Class I recommendation. However, recent randomized controlled trials have demonstrated that high-risk patients with complex coronary artery disease or high-risk clinical conditions still experience a continuous increase in adverse cardiovascular events despite optimal secondary prevention. This underscores the need for an optimized surveillance strategy to improve long-term prognosis.

Despite the emphasis on GDMT and secondary prevention in current guidelines, the most effective surveillance strategy after PCI remains uncertain. Existing recommendations primarily address secondary prevention and provide only limited guidance on surveillance for patients with previous coronary revascularization. Based on multiple randomized controlled trials, current guidelines do not recommend routine non-invasive stress testing or coronary CT angiography (CCTA) in asymptomatic patients receiving optimized GDMT (Class III, Level of Evidence B-R). However, this recommendation lacks direct evidence evaluating CCTA as a surveillance strategy after PCI. In patients with prior coronary revascularization, CCTA is currently recommended for assessing bypass graft or stent patency only in symptomatic patients (Class IIa), with limited supporting evidence (Level of Evidence B in ESC guidelines and Level of Evidence B-NR in ACC/AHA guidelines).

Notably, the SCOT-HEART trial demonstrated that a CCTA-based treatment strategy was superior to standard care, which relied on clinical and functional assessment along with as-needed non-invasive stress testing, in reducing a composite outcome of coronary heart disease death and non-fatal myocardial infarction. This suggests that a surveillance strategy incorporating CCTA may lead to improved subsequent management decisions, such as preemptive ischemia-driven revascularization or intensified medical therapy, potentially reducing ischemic cardiovascular events and mortality compared to standard guideline-recommended care.

To address this critical gap in clinical practice, we designed the Smart Angioplasty Research Team-Coronary CT Angiography versus Standard Care as Follow-up Strategies in High-Risk Patients after PCI (SMART-CARE) trial. This study aims to evaluate the impact of a CCTA-based surveillance strategy on clinical outcomes compared with standard guideline-directed follow-up in high-risk patients who have undergone PCI.

ELIGIBILITY:
Inclusion Criteria:

① Patients aged 19 years old

② Patients who underwent successful PCI with one or more contemporary drug-eluting stents (stent diameter ≥3mm) or drug-coated balloons.

③ Patients must have at least one of the following criteria of complex coronary artery lesions or high-risk clinical characteristics:

A. Complex coronary artery lesions:

i. True bifurcation lesion (Medina 1,1,1/1,0,1/0,1,1) with side branch ≥2.5mm size ii. Chronic total occlusion (≥3 months) as target lesion iii. PCI for unprotected left main (LM) disease (LM ostium, body, distal LM bifurcation including non-true bifurcation) iv. Long coronary lesions (used stents or drug-coated balloons ≥38 mm in length) v. Multi-vessel PCI (≥2 major epicardial coronary arteries treated at one PCI session) vi. Multiple devices needed (≥3 more stents or drug-coated balloons per patient) vii. In-stent restenosis lesion as target lesion viii. Severely calcified lesion (encircling calcium in angiography) ix. Left anterior descending (LAD), left circumflex artery (LCX), and right coronary artery (RCA) ostial lesion

B. High-risk clinical characteristics:

i. Acute myocardial infarction (ST-elevation myocardial infarction [MI] or non-ST-elevation MI) with or without cardiogenic shock (SCAI Classification ≥C) at presentation ii. Diabetes mellitus which requires medical treatment (oral hypoglycemic agents or insulin) iii. End-stage renal disease under dialysis iv. Combined vascular disease other than coronary artery disease

1. Peripheral artery occlusive disease which is defined as A. Previous aorto-femoral bypass surgery, limb bypass surgery, or percutaneous transluminal angioplasty revascularization of the iliac, or infra-inguinal arteries, or B. Previous limb or foot amputation for arterial vascular disease, or C. History of intermittent claudication and one or more of the following: 1) An ankle/arm blood pressure (BP) ratio < 0.90, or 2) Significant peripheral artery stenosis (≥50%) documented by angiography, or by duplex ultrasound, or D. Previous carotid revascularization or asymptomatic carotid artery stenosis ≥50% as diagnosed by duplex ultrasound or angiography.
2. Thoracoabdominal aortic disease which is defined as A. Documented thoracoabdominal aortic aneurysm by duplex ultrasound, angiography, or computed tomography angiography B. Previous endovascular or surgical treatment for thoracoabdominal aortic aneurysm

   ④ Subject who can verbally confirm understandings of risks, benefits and surveillance strategy alternatives of receiving CCTA and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

   Exclusion Criteria:

   ① Advanced chronic kidney disease (Creatinine clearance <30 ml/min/1.73 m2) not on dialysis
   * Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)

     * Pregnancy or breast feeding ④ Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment) ⑤ Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first event of major adverse cardiac events (MACE) | 2 years after the last patient enrollment
  MACE is a composite of death, non-fatal myocardial infarction (MI), hospitalization for acute coronary syndrome leading to an urgent revascularization, or stent thrombosis

SECONDARY OUTCOMES:
All-cause death | 2 years after the last patient enrollment
  All-cause death
Cardiac death | 2 years after the last patient enrollment
  Cardiac death
Non-fatal MI | 2 years after the last patient enrollment
  Non-fatal MI, defined by Forth Universal definition of MI
Spontaneous MI | 2 years after the last patient enrollment
  Spontaneous MI, defined by Forth Universal definition of MI
Procedure-related MI (during follow-up period from invasive procedure) | 2 years after the last patient enrollment
  Procedure-related MI (during follow-up period from invasive procedure), defined by Fourth Universal definition of MI
Hospitalization for acute coronary syndrome leading to an urgent revascularization | 2 years after the last patient enrollment
  Hospitalization for acute coronary syndrome is defined as a clinical event in which the final diagnosis during unplanned hospitalization is acute coronary syndrome including spontaneous myocardial infarction or unstable angina.
Unplanned revascularization (clinically-driven) | 2 years after the last patient enrollment
  All revascularization events will be adjudicated as either clinically-driven or non-clinically-driven. Revascularization will be considered clinically-driven if the diameter stenosis of the revascularized coronary segment is ≥50% by QCA and any of the following criteria for ischemia are met:
  * A positive functional study corresponding to the area served by the target lesion; or
    * Ischemic ECG changes at rest in a distribution consistent with the target vessel; or
      * Typical ischemic symptoms referable to the target lesion; or ④ positive invasive physiologic test (fractional flow reserve ≤0.80 or instantaneous wave-free ratio ≤0.89); or ⑤ presence of stenosis with ≥70% diameter stenosis, even in the absence of other criteria Unplanned revascularization refers to revascularization not planned after initial assessments with invasive coronary angiography or non-invasive stress testing, depending on the allocated group, but performed due to clinical circumstances.
Definite stent thrombosis | 2 years after the last patient enrollment
  Definite stent thrombosis, defined by Academic Research Consortium (ARC) II consensus
Rate of invasive coronary angiography during follow-up | 2 years after the last patient enrollment
  Rate of invasive coronary angiography (with or without showing restenosis or obstructive CAD) during follow-up.
  Angiographic restenosis was defined as a stenosis of at least 50 percent of the minimal luminal diameter in the target-lesion at invasive coronary angiography during follow-up. Obstructive or no obstructive coronary artery disease at invasive coronary angiography is defined as a visually estimated presence or absence of stenosis of 50% or more, as interpreted by the study-site staff, in any major epicardial vessel, including side branches of at least 2.5 mm in diameter.
Rate of revascularization by PCI or CABG during follow-up | 2 years after the last patient enrollment
  Rate of revascularization by PCI or CABG during follow-up
Procedure-related complications from invasive procedure during follow-up | 2 years after the last patient enrollment
  Procedure-related complications from invasive procedure during follow-up
Cerebrovascular accidents | 2 years after the last patient enrollment
  Cerebrovascular accidents (ischemic or hemorrhagic)
Contrast-induced nephropathy or contrast-associated hypersensitivity reaction | 2 years after the last patient enrollment
  Contrast-induced nephropathy, defined as an increase in serum creatinine of ≥0.5mg/dL or ≥25% from baseline within 48-72 hours after contrast agent exposure or contrast-associated hypersensitivity reaction
Total medical cost | 2 years after the last patient enrollment
  Total medical cost
A composite of death or non-fatal MI | 2 years after the last patient enrollment
  A composite of death or non-fatal MI

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (22):
- South Korea (22):
  - SoonChunHyang University Hospital Bucheon, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Chonnam National University Medical School, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Inje University College of Medicine, Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Kwandong University Intl. ST. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Chung-Ang University College of Medicine, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, College of Medicine, Hanyang University, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Kuro Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.